CLINICAL TRIAL: NCT06693661
Title: Improving Access to Nephrology Treatment and Care Among Patients at Greatest Risk for Kidney Failure
Brief Title: Collaborative Learning to Achieve Refined Interventions for Emory: Kidney Disease
Acronym: CLARIFy-KD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); James T. Laney School of Graduate Studies (Unknown)
Responsible Party: Principal Investigator, Kimberly R Jacob Arriola, Vice Provost for Graduate Studies, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY00007938; 1U01DK137269 (NIH); 2025P008750 (Other: Emory IRB)
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Kidney Diseases
Keywords: African American; Health Disparities; Chronic Care Model (CCM); Kidney Health Coach (KHC)
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Kidney Health Coaching (Other): Participants will receive patient-centered health coaching delivered by two full-time kidney health coaches for six months.
  Interventions: Other: Kidney Health Coaching
- Control: Usual Care (Other): Participants will receive the usual care based on where patients are identified (Emergency Room- ER, Primary Care, Hospital Discharge, Primary Care, or Nephrology)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Kidney Health Coaching — The intervention entails support from a KHC that includes:
  * An initial rapport-building call
  * Ongoing telephone support at least twice a month for six months
  * Meeting the patient at all in-person clinic appointments
  * Documenting interactions in the EMR using a customized platform
  Telephone support begins with a social determinants of health (SDoH) screening tool to identify barriers and facilitators to CKD self-management and appointment adherence. This tool provides access to local resources based on the patient's ZIP code. Subsequent calls will follow up on resource usage, review CKD educational materials and treatment options, complete the Decision Aid for Renal Therapy tool, and facilitate communication through the patient portal. Each call will start with specific goals (e.g., review National Kidney Foundation CKD materials) and conclude with goals for the next session.
  Other Names: KHC Protocol
  Arms: Intervention: Kidney Health Coaching
Other: Usual Care — ER Discharge (d/c): Participants may receive consultations and support from Care Management in the ER, such as transportation or medication assistance. Follow-up by a social worker varies post-discharge.
  Hospital d/c: All hospitalized patients are assessed by the care management team to identify psychosocial needs and begin discharge planning, which may include follow-up appointments and resources. High-risk patients receive additional follow-up from a care transitions coordinator for 30 days post-discharge.
  Primary Care: Patients in primary care clinics have access to various support services. Those recently hospitalized or identified as high-risk receive care coordination from social workers. Internal referrals are managed by referral coordinators, while external referrals come from clinic staff. Discharge information is provided after visits.
  Nephrology: There are no coordinated support services for chronic kidney disease (CKD) patients receiving nephrology care.
  Other Names: Control
  Arms: Control: Usual Care

SUMMARY:
Through the use of community-engaged processes, this project seeks to develop and implement clinical decision support (CDS) and a kidney health coaching (KHC) intervention. The CDS seeks to streamline workflows to effectively screen, identify, and link to care for those patients with advanced chronic kidney disease (CKD).

The overall project goals are to 1.) Design and conduct community-engaged clinical trials to test new interventions that dismantle the systemic factors that contribute to kidney health disparities. 2.) Foster research collaborations between investigators, people living with kidney disease, community-based organizations, and other key stakeholders.

Researchers aim to assess whether the KHC intervention is effective at delaying the transition to kidney replacement therapy (KRT) and central venous catheter use or death.

DETAILED DESCRIPTION:
This study has two Aims. In Aim 1, the research team will develop and implement multi-level, multi-component interventions across primary care and acute care access points, nephrology, and dialysis care using the Chronic Care Model as an organizing framework.

Aim 1: Implement multi-level, multi-component interventions across primary care and acute care access points, nephrology, and dialysis care using the Chronic Care Model as an organizing framework. The research team will deliver patient-centered kidney health coaching, with full-time kidney health coaches (KHC). They must have lived experience with chronic kidney disease (CKD) and will be selected for certain personality characteristics. The KHCs will undergo training to deliver patient support that aligns with 4 constructs of the Chronic Care Model: Clinical information systems, Patient self-management, and treatment decision-making support, Delivery system redesign, and Community resources. Participants enrolled in the intervention will receive 6-months of kidney health coaching. Those eligible for participation will be invited to participate and undergo the informed consent process via telephone. Next, study staff will administer the baseline assessment via telephone interview for those who consent.

Aim 2: Using a 2-group randomized controlled trial, determine the effectiveness of the interventions on primary outcomes analyzed at the level of patients (i.e., referral to nephrology and preemptive transplant, uptake of home hemodialysis).

ELIGIBILITY:
Inclusion Criteria:

* Identifies as African American or Black;
* Two estimated glomerular filtration rates (eGFRs) < 29 separated by at least 90 days but within the past 2 years or a Kidney Failure Risk Equation (KFRE) score of 10% or greater likelihood of kidney failure within the next 2 years;
* Had an encounter at Emory University Hospital-Midtown through an ambulatory visit or inpatient stay (i.e., ER or hospital visit within the previous 2 months
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Currently on dialysis
* currently receiving hospice care or other types of conservative management for terminal illness
* Currently on waitlist, or referred for/or completed a transplant evaluation visit within the past 2 years
* Kidney or another solid organ transplant
* Active cancer treatment
* Non-English speaking
* Participating in another treatment or intervention study at the time of enrollment
* Currently pregnant or planning to become pregnant at the time of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Time-to-Kidney Replacement Therapy w/Central Venous Catheter | Throughout study participation up to 12 months
  Composite measure of time to transition to Kidney Replacement Therapy (KRT) using a central venous catheter (CVC) over the course of the study period
Time-to-death | Throughout study participation up to 12 months
  Composite measure of time to death over the course of the study period. A record of death in the electronic medical record (EMR), and the date of death will be recorded. If the data is not available in EMR, national death statistics will be checked, and the patient's family will be asked.

SECONDARY OUTCOMES:
Time to progression to end stage kidney disease (ESKD) | Throughout study participation up to 12 months
  Composite measure of time to ESKD diagnosis over the course of the study period. Progression to ESKD will be analyzed using monthly data collected from the EMR, capturing each participant's progression characterized by a significant loss of kidney function (defined as a glomerular filtration rate (GFR) of less than 15 mL/min) requiring KRT. Time to event will be calculated for all participants at the end of the follow-up period.
Time-to-optimal Kidney Replacement Therapy (KRT) referral | Throughout study participation up to 12 months
  Composite measure of time to referral for optimal KRT start over the course of the study. This includes referral for vascular surgery, preemptive kidney transplant evaluation, and/or home dialysis initiation. Data will be collected monthly from the EMR.
Number of participants who transition-to-Kidney Replacement Therapy w/Central Venous Catheter | Throughout study participation up to 12 months
  Number of participants who transitioned to Kidney Replacement Therapy (KRT) with the use of a central venous catheter (CVC) during the course of the study.
Mortality rate | Throughout study participation up to 12 months
  Mortality during study participation.
Proportion of nephrology appointment attendance | Throughout study participation up to 12 months
  Continuous measure of nephrology appointment adherence measured as the ratio of # appointments attended to # appointments scheduled during the course of the study. At the end of the follow-up period for all participants, the researchers will calculate the proportion of appointments attended as a measure of appointment adherence. This will be captured from the Emory Healthcare appointment-keeping system.
CKD Symptom Burden | Baseline, 6 months and 12 months
  Self-reported occurrence of physical and emotional symptoms commonly experienced in individuals with CKD. Participants will complete a 29-item CKD Symptom Burden questionnaire that captures the frequency at which patients experience symptoms. Response options are on a 4-point scale (0 'never' to 4 'every day'). The summed total score ranges from 0 to 29. The greater the frequency of symptoms, the poorer the health-related and self-perceived quality of life.
Quality of Life Scale | Baseline, 6 months and 12 months
  Participants will complete a 10-item phone survey that assesses their perceived quality of life. Responses are recorded on a 5-point scale, with total scores ranging from 10 to 50; higher scores indicate better self-reported health-related quality of life.
Patient activation Score | Baseline, 6 months and 12 months
  Patient activation will be measured using the Patient Activation Measure (PAM), completed by phone. PAM is a validated self-reported questionnaire designed to assess an individual's knowledge, skills, and confidence in managing their well-being. It captures participants' agreement with 22 statements regarding their self-efficacy in maintaining health, measured on a scale from "Strongly Disagree" to "Strongly Agree." The response options are on a 4-point scale. Scores range from 0 to 100, with higher scores indicating greater activation.
Decisional conflict scale | Baseline, 6 months and 12 months
  Decisional conflict will be measured using the Decisional Conflict Scale (DCS). The DCS measures personal perceptions of uncertainty in choosing options. The survey will be conducted over the phone to capture the level of agreement a participant has with 16 statements regarding their ability to make an informed decision, measured on a scale from "Strongly Disagree" to "Strongly Agree." This information will be collected at baseline, 6, and 12 months. The response options are on a 5-point scale. Scores can range from 16 to 70. Higher Scores indicate higher decisional conflicts.
Medical Mistrust Organization Score | Baseline, 6 months and 12 months
  Medical mistrust organization will be measured using the Medical Mistrust Index adapted to address general mistrust of healthcare providers. Participants will answer the questions over the phone. Questions will capture their level of agreement with seven statements regarding healthcare organizations. Responses are measured on a 4-point scale, ranging from "Strongly Disagree" to "Strongly Agree". Scores can range from 7 to 28.
CKD treatment Knowledge | Baseline, 6 months and 12 months
  To measure participants' CKD treatment knowledge, they will complete a 9-item yes/no questionnaire over the phone. The research team will count the number of correct responses, resulting in a score ranging from 0 to 9.
Rotterdam Renal Replacement Knowledge test | Baseline, 6 months and 12 months
  KRT knowledge will be measured using the Rotterdam Renal Replacement Knowledge test. Participants will complete the 21-item test over the phone, assessing their understanding of renal replacement therapy. The research team will count the correct responses, allowing scores to range from 0 to 21. Higher scores suggest a better understanding of KRT, indicating preparedness to make informed decisions about treatment options.
Shared Decision-Making Score | Baseline, 6 months and 12 months
  Shared decision-making will be measured using the Shared Decision-Making Q-9. Participants will respond by phone to 16 statements regarding their ability to make informed decisions, using a 5-point scale from "Strongly Disagree" to "Strongly Agree." Scores will range from 16 to 80.
  Low Score (16-40): Indicates poor shared decision-making, suggesting the patient may feel uninformed or not involved in their care.
  Moderate Score (41-60): Reflects a moderate level of shared decision-making, indicating some collaboration occurs but that improvements are needed.
  High Score (61-80): Suggests strong shared decision-making, where patients feel well-informed and actively involved in their healthcare decisions.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly R Jacob Arriola, PhD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigator will share individual de-identified data that supports statistical analysis
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following the completion of the study.
Access Criteria: Through the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Data Repository.
URL: https://repository.niddk.nih.gov/home